CLINICAL TRIAL: NCT01341847
Title: The Water Method Colonoscopy in Routine Unsedated Colonoscopy Examinations : A Randomized Controlled Trial(RCT) in Diagnostic Cases in Indonesian Patients
Brief Title: The Water Method Colonoscopy in Routine Unsedated Colonoscopy Examinations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, PUTUT BAYUPURNAMA, MD, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PB-63
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Colonoscopy Diagnostic Techniques and Procedures

ARMS (2):
- Water method colonoscopy (Active Comparator): This technique allow only water infusion (air pump is turned off) through the adaptor on the biopsy channel of the colonoscope during insertion since the scope is inserted into the anus until reach the cecum. Water will be infused as needed under endoscopist judgement through the adaptor on biopsy channel with endoscopic washer pump. The usual air insufflation will be used during colonoscope withdrawal to facilitate mucosal examination and perform any other intervention, such as biopsy
  Interventions: Procedure: water method colonoscopy
- air method colonoscopy (Other): This technique only use usual air insufflation technique during colonoscope insertion and shortening maneuvers.
  Interventions: Procedure: air method colonoscopy

INTERVENTIONS:
Procedure: water method colonoscopy — This technique allow only water infusion (air pump is turned off) through the adaptor on the biopsy channel of colonoscope during insertion since the scope is inserted into the anus until reach the cecum.
  Arms: Water method colonoscopy
Procedure: air method colonoscopy — This technique only use usual air insufflation technique during colonoscope insertion and shortening maneuvers.
  Arms: air method colonoscopy

SUMMARY:
Aim of the Study :

This study will compare the colonoscopy examination between the air method (air insufflation) and water method (water infusion) in unsedated patients with indication (symptoms and signs based) of colonoscopy examination. This study is based on earlier study which showed that water method had better results in reducing abdominal pain, caecal intubation and patients willingness to repeat colonoscopy examination than air method.

Background:

Colonoscopy examination is an important method to examine and establish the diagnosis of various diseases in the colon. Colonoscopy is successful when the tip of the scope reach the cecum and observe the caecal valve and/ or appendix orifice. This examination can be performed unsedated or under sedation (conscious sedation or deep sedation/general anaesthesia). The main disadvantage of unsedated colonoscopy method is the abdominal discomfort or pain during examination that may make patient distress and hemodynamically unstable and possibly stoppage of the examination before reach the cecum, but the severity of abdominal symptoms is vary from patient to patient. Many efforts have been tried to reduce the abdominal discomfort during examination. This unsedated method with air insufflation is our hospital standard method for colonoscopy examination since early 1980s, and less than 1% of patients were colonoscopied with conscious or deep sedation. Our study showed the success rate of this standard unsedated method was about 82%. The advantage of this method is inexpensive (feasible for most of people in developing country like us), patient may be examined ambulatory without escort, may back to work as soon as the examination is finished. Studies showed that replace the air insufflation with water infusion into colon since the beginning of the examination increased the success rate of caecal intubation and reduced the abdominal pain symptoms during colonoscopy examination(1). Sedation or general anaesthesia may increase the success rate of colonoscopy examination but it is costly, and may increase the adverse event especially in the elderly or patients with significance cardiopulmonary problems.

Research Design and Methods:

Eligible patients in the hospital clinics or wards will be offered to follow unsedated colonoscopy examination. The principle investigator (PI) will explain the study, the colonoscopy procedure , the various symptoms that may be felt during examination, the possible adverse event and medical effort to prevent it. Patient who sign the informed consent will be included in the study.

Methods on the day of exam. Enrolled patients will be sent to the endoscopy room and colonoscopy will be performed by the principle investigator. Patient lie on the left lateral position with right hip and knee flexed and left leg straight. When the PI about to start the single-handed colonoscopy examination, the blinded observer open the sealed envelops with the code enclosed. A standard colonoscope will be inserted. Patient may be ordered to change the position and or abdominal compression may be applied by nurse to aid the colonoscope advancement. Oximetry, cardiac rhythm and blood pressure will be monitored during examination. Blinding will not be performed in this study because of the feeling of water or air effect inside the colon can be differentiated by the patient so that in our opinion it actually can not be blinded..The control method includes usual air insufflation during insertion and shortening maneuvers. The study method includes only water infusion (air pump is turned off) through the colonoscope during insertion since the scope is inserted into the anus until reach the cecum. Water will be infused as needed under endoscopist judgement through the adaptor on biopsy channel with endoscopic washer pump. The usual air insufflation will be used during colonoscope withdrawal to facilitate mucosal examination and perform any other intervention, such as biopsy. Hypothesis testing: The unsedated colonoscopy with natural temperature water infusion minimize the pain symptoms than unsedated colonoscopy with usual air insufflation.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years old with indication for colonoscopy, such as chronic diarrhea, chronic constipation, hematochezia, chronic lower abdominal pain, positive fecal occult blood test, and other change of bowel habit symptoms indicative for colonoscopy examination

Exclusion Criteria:

* Patients refuse to participate
* Patient with obstructive lesion in the colon distal of the cecum,
* Patients with experienced of colon resection, hemodynamically unstable,severe cardiac disorders (such as acute myocardial infarction,unstable angina,malignant arrhythmia, and moderate to severe congestive heart failure,
* Patients with fecal obstruction (whatever the cause) so that impossible to pass the scope through the obstructed segment;
* Patients with communication problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Abdominal discomfort score | one year
  The level of abdominal discomfort experienced by the patient during the colonoscopy examination and reported to a blinded observer shortly before discharge (5 to 10 minutes after colonoscopy) will be measured on a linier visual analog scale :0=none, 10= most severe

SECONDARY OUTCOMES:
Cecal Intubation | one year
  Touching the tip of the colonoscope to the cecum with visualization of the ileocecal valve and/or appendix orifice

CONTACTS AND LOCATIONS:
Overall Officials: Putut Bayupurnama, MD, Principal Investigator — Division of Gastroenterology and Hepatology, Department of Internal Medicine, Faculty of Medicine, Gadjah Mada University/Sardjito General Hospital, Yogyakarta, Indonesia
Locations (1):
- Endoscopy Room of Dr Sardjito General Hospital, Yogyakarta, Special Province of Yogyakarta, Indonesia